CLINICAL TRIAL: NCT00487435
Title: Open-Label Extension, Single-Arm, Flexible-Dosing, Phase 3 Trial With CG5503 Extended-Release (ER) in Patients With Moderate to Severe Chronic Pain
Brief Title: An Open-label Extension Study With Flexible Dosing of Extended-release (ER) Tapentadol (CG5503) to Treat Patients With Moderate to Severe Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013567; R331333PAI3010; KF18
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Results first posted 2010-07-23 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Pain; Osteoarthritis; Low Back Pain
Keywords: CG5503; Tapentadol; chronic non-malignant pain; osteoarthritis; lower back pain; analgesic; opioid
MeSH Terms: conditions — Pain; Osteoarthritis; Low Back Pain | interventions — Tapentadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): Tapentadol (CG5503) Extended Release (ER) 100 150 200 250 mg oral tablet twice daily for 52 weeks
  Interventions: Drug: Tapentadol (CG5503) Extended Release (ER)

INTERVENTIONS:
Drug: Tapentadol (CG5503) Extended Release (ER) — 100, 150, 200, 250 mg oral tablet twice daily for 52 weeks

SUMMARY:
The purpose of the study is to assess the long-term safety profile of Tapentadol (CG5503) extended release (ER) at dosages ranging from 100 to 250 mg twice a day in treating patients with moderate to severe chronic pain over a period of 1 year. The study will also assess dosage requirements over the long term; characterize adverse events and tolerability, sleep quality, and potential symptoms of withdrawal; characterize pain intensity scores and overall impression of change; and characterize patient-related health outcomes.

DETAILED DESCRIPTION:
All patients who complete the Phase 3 pivotal trials in osteoarthritis (R331333-PAI-3008; KF5503/11) and low back pain (R331333-PAI-3011; KF5503/23) and the Phase 3 safety trial in the non-European sites (R331333-PAI-3007; KF5503/24) will be allowed to continue participation in the program by entering this trial. The trial will consist of three periods (screening, open-label treatment period, and follow-up). In the open-label treatment/maintenance period (1 year), those patients in the safety trial R331333-PAI-3007 (KF5503/24) taking open-label Tapentadol (CG5503) extended release (ER) will continue the dosage they were taking without undergoing titration. All other patients will be titrated to the minimum therapeutic dosage of Tapentadol (CG5503) extended release (ER) over 1 week. The lowest therapeutic dose allowed in the study is 100 mg twice daily, and the maximum upper dosage of Tapentadol (CG5503) extended release (ER) base is 250 mg twice daily. Downward titration (not below the minimum therapeutic dose of 100 mg twice daily) is permitted at any time using the same decrements without any time restriction. Dosages will be assessed at the scheduled (and unscheduled, if any) visits and adjustment under investigator supervision will be made as necessary. Dosage adjustments should be kept to a minimum. Intake of paracetamol/acetaminophen two 500 mg tablets daily is permitted during the titration week, and during the remainder of the open-label treatment/maintenance period up to a maximum of 7 consecutive days but no more than 14 out of 30 days. Following Week 4, all visits will be scheduled at 4-week intervals, through Week 52. The end-of-treatment visit at Week 52 will include both safety and efficacy assessments. Patients will return to the site for a follow-up visit approximately 4 days after their last dose of Tapentadol (CG5503) extended release (ER) for final safety evaluations and completion of the opioid withdrawal assessments (clinical opioid withdrawal scale, or COWS, and subjective opioid withdrawal scale, or SOWS). Patients experiencing withdrawal symptoms prior to the follow-up visit may telephone and request to be seen sooner. Additionally, the research staff at the site will telephone subjects approximately 10 to 14 days after the last dose of Tapentadol (CG5503) extended release (ER) to inquire if any adverse events have occurred since the previous visit. Tapentadol (CG5503) extended release (ER): 50, 100, 150, 200, and 250 mg orally, taken twice daily (morning and evening) for a maximum duration of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Non-lactating female subjects (Sexually active women must be postmenopausal, surgically sterile, or practicing an effective method of birth control [e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, contraceptive patch, male partner sterilization] before entry and throughout the trial. Female patients of childbearing potential must have a negative pregnancy test at screening.)
* Completion of the expected double-blind treatment period of the pivotal Tapentadol (CG5503) Phase 3 trials in osteoarthritis (R331333-PAI-3008, KF5503/11) or low back pain (R331333-PAI-3011, KF5503/23), or completion of the 1-year treatment period of the safety CG5503 Phase 3 trial in the non-European sites (R331333-PAI-3007, KF5503/24)
* Must be willing to take Tapentadol (CG5503) extended release (ER) and the rescue medication supplied for the duration of the trial

Exclusion Criteria:

* History of alcohol and/or drug abuse, life-long history of seizure disorder or epilepsy, any of the following within the past year: mild/moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm
* Severe traumatic brain injury within the past 15 years
* Uncontrolled hypertension (repeated systolic blood pressure >160 mmHg or diastolic blood pressure >95 mmHg)
* Severely impaired renal function
* Moderately or severely impaired hepatic function
* Patients taking neuroleptics, monoamine oxidase inhibitors, or tricyclic antidepressants within 14 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1166 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (148):
- United States (118):
  - Birmingham, Alabama
  - Hoover, Alabama
  - Mobile, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Carmichael, California
  - Encinitas, California
  - Fresno, California
  - Huntington Park, California
  - Laguna Hills, California
  - Los Gatos, California
  - Pico Rivera, California
  - Pismo Beach, California
  - Sacramento, California
  - San Diego, California
  - Upland, California
  - Westlake Village, California
  - Stamford, Connecticut
  - Trumbull, Connecticut
  - Chiefland, Florida
  - Clearwater, Florida
  - Fort Myers, Florida
  - Hallandale, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Oldsmar, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - Port Orange, Florida
  - Sarasota, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Athens, Georgia
  - Augusta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Perry, Georgia
  - Suwanee, Georgia
  - Woodstock, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Avon, Indiana
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Valparaiso, Indiana
  - West Des Moines, Iowa
  - Overland Park, Kansas
  - Prairie Village, Kansas
  - Topeka, Kansas
  - Madisonville, Kentucky
  - Baton Rouge, Louisiana
  - Lake Charles, Louisiana
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Columbia, Maryland
  - Owings Mills, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Brighton, Massachusetts
  - Fall River, Massachusetts
  - North Dartmouth, Massachusetts
  - Wellesley Hills, Massachusetts
  - West Yarmouth, Massachusetts
  - East Lansing, Michigan
  - Grand Blanc, Michigan
  - Kalamazoo, Michigan
  - Troy, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Cherry Hill, New Jersey
  - Albuquerque, New Mexico
  - Mamaroneck, New York
  - New York, New York
  - Williamsville, New York
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Kettering, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Allentown, Pennsylvania
  - Chester, Pennsylvania
  - Duncansville, Pennsylvania
  - Morrisville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
  - Prosperity, South Carolina
  - Sioux Falls, South Dakota
  - Clarksville, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Hurst, Texas
  - Lubbock, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Danville, Virginia
  - Roanoke, Virginia
  - Virginia Beach, Virginia
  - Bellevue, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin
- Australia (4):
  - Adelaide
  - Melbourne
  - Newcastle
  - Woodville North
- Canada (23):
  - Chilliwack, British Columbia
  - Kelowna, British Columbia
  - Penticton, British Columbia
  - Vancouver, British Columbia
  - St. John's, Newfoundland and Labrador
  - Ajax, Ontario
  - Brampton, Ontario
  - Greater Sudbury, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Markham, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Vancouver, Ontario
  - Charlottetown, Prince Edward Island
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Saint Romuald, Quebec
  - Sherbrooke, Quebec
  - Saskatoon, Saskatchewan
  - Halifax
- New Zealand (3):
  - Christchurch
  - Tauranga
  - Wellington

REFERENCES:
- [Derived] Buynak R, Rappaport SA, Rod K, Arsenault P, Heisig F, Rauschkolb C, Etropolski M. Long-term Safety and Efficacy of Tapentadol Extended Release Following up to 2 Years of Treatment in Patients With Moderate to Severe, Chronic Pain: Results of an Open-label Extension Trial. Clin Ther. 2015 Nov 1;37(11):2420-38. doi: 10.1016/j.clinthera.2015.08.014. Epub 2015 Oct 1. PMID 26428249
- See also: An open-label extension study with flexible dosing of extended-release (ER) Tapentadol (CG5503) to treat patients with moderate to severe chronic pain — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=70&filename=CR013567_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this out-patient, multicenter study occurred between 4 June 2007 and 29 June 2009.
Groups:
- Tapentadol (CG5503) Extended Release (ER): Tapentadol (CG5503) extended release (ER) 100 to 250mg oral tablet twice daily (BID) for up to one year
Period: Overall Study
Arm/Group | Tapentadol (CG5503) Extended Release (ER)
Started | 1154 (Patients who received at least one dose of Tapentadol (CG5503) Extended Release (ER))
Completed | 669
Not Completed | 485
Not completed — Adverse Event | 146
Not completed — Death | 2
Not completed — Lack of Efficacy | 33
Not completed — Lost to Follow-up | 54
Not completed — Pregnancy | 2
Not completed — Withdrawal by Subject | 132
Not completed — Resolution Of Pain | 1
Not completed — Study Medication Non-Compliant | 32
Not completed — Other | 83

BASELINE CHARACTERISTICS:
Arm/Group | Tapentadol (CG5503) Extended Release (ER)
Number analyzed (Participants) | 1154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 954
  >=65 years | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 668
  Male | 486
Region Enroll [Number; unit: participants]
  Australia | 15
  Canada | 178
  New Zealand | 10
  United States of America | 951

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAE)
Description: The number of subjects who reported a TEAE during the treatment period. TEAE was defined as any adverse event that started or worsened on or after the start of the study medication and up to 3 days after the discontinuation of the study medication.
Time Frame: 52 weeks
Population: Safety analysis set (All randomized subjects who took at least one dose of study medication).
Measure: Number; unit: participants
Arm/Group | Tapentadol (CG5503) Extended Release (ER)
Number analyzed (Participants) | 1154
participants | 907

2. Secondary Outcome: Change From Baseline in Average Pain Intensity Scores at Week 52 Using the Numerical Rating Scale (NRS)
Description: The subjects indicated the average level of pain experienced, at each study visit, over the previous 24 hours on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Baseline, 52 weeks
Population: observed cases
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Tapentadol (CG5503) Extended Release (ER)
Number analyzed (Participants) | 711
Scores on a Scale | -0.26 (2.129)

ADVERSE EVENTS:
Description: Only subjects who had at least one of the TEAEs listed in the Other (non Serious) AE table are included in the Total no. subjects with Non-Serious Adverse Events.
Arm/Group | Tapentadol (CG5503) Extended Release (ER)
Serious Adverse Events (participants affected / at risk) | 84/1154
Other Adverse Events (participants affected / at risk) | 659/1154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (CG5503) Extended Release (ER) (N=1154)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall mass (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cor pulmonale (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Chest pain (General disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Drug withdrawal syndrome (General disorders) | 1
Hernia obstructive (General disorders) | 1
Influenza like illness (General disorders) | 1
Gastroenteritis viral (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Bursitis infective (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Mastitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 3
Abdominal injury (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Coma (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Altered state of consciousness (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Intraventricular haemorrhage (Nervous system disorders) | 1
Suicidal ideation (Psychiatric disorders) | 2
Withdrawal syndrome (Psychiatric disorders) | 2
Completed suicide (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Suicidal behaviour (Psychiatric disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Colitis ischaemic (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Cystocele (Reproductive system and breast disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Lipase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Colectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (CG5503) Extended Release (ER) (N=1154)
Nausea (Gastrointestinal disorders) | 135
Constipation (Gastrointestinal disorders) | 128
Diarrhoea (Gastrointestinal disorders) | 110
Vomiting (Gastrointestinal disorders) | 71
Headache (Nervous system disorders) | 151
Dizziness (Nervous system disorders) | 98
Somnolence (Nervous system disorders) | 61
Nasopharyngitis (Infections and infestations) | 77
Upper respiratory tract infection (Infections and infestations) | 71
Sinusitis (Infections and infestations) | 63
Urinary tract infection (Infections and infestations) | 63
Insomnia (Psychiatric disorders) | 100
Anxiety (Psychiatric disorders) | 61
Fatigue (General disorders) | 77
Arthralgia (Musculoskeletal and connective tissue disorders) | 63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less